CLINICAL TRIAL: NCT03932136
Title: Decreasing Risk of Psychosis by Sulforaphane: Study Protocol for a Randomized, Double-blind, Placebo-controlled, Clinical Multicenter Trial (DROPS Trial)
Brief Title: Decreasing Risk of Psychosis by Sulforaphane (DROPS Trial)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Xuhui District Mental Health Center (Unknown); Shanghai Pudong Nanhui Mental Health Center (Unknown); Suzhou Psychiatric Hospital (Other); Second Xiangya Hospital of Central South University (Other); Guangzhou Psychiatric Hospital (Other Government); Shenzhen Fushan Biotech Co., Ltd. (Unknown); Tianjin Anding Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Shenzhen Kangning Hospital (Other)
Responsible Party: Principal Investigator, Jijun Wang, Professor, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 03
Record Dates: First submitted 2019-04-23; First posted 2019-04-30 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Clinical High Risk Syndrome of Psychosis
MeSH Terms: interventions — sulforaphane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SFN group (Active Comparator): The intervention duration with SFN tablet is 52 consecutive weeks. The dosage is six active tablets (411 μmol GR) per day.
  Interventions: Dietary Supplement: Sulforaphane
- Placebo group (Placebo Comparator): The intervention duration with placebo tablet is 52 consecutive weeks. The placebo group will be given six placebo tablets per day.
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Dietary Supplement: Sulforaphane — Sulforaphane (SFN) is a natural compound extracts from cruciferous vegetables, especially broccoli, with cytoprotective, anti-inflammatory, and antioxidant effects.
  Other Names: ZHIYINGUOSU
  Arms: SFN group
Combination Product: Placebo — The placebo is safe, with no therapeutical effect, and has same appearance and similar smell and taste with active tablet.
  Arms: Placebo group

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multi-centre trial. A total of 300 CHR subjects will be identified in the course of face-to-face interviews using the Structured Interview for Prodromal Syndromes. All participants will be randomly allocated to SFN group (n = 150) or placebo group (n = 150). The study duration includes an intervention for 52 consecutive weeks, and additional 1-year follow-up. The primary outcome is 2-year conversion rate of psychosis. Secondary outcomes include 1-year conversion rate of psychosis, the severity and duration of prodromal symptoms, predictive risk of psychosis conversion, neurocognitive functioning and peripheral blood biomarkers of inflammation, oxidative stress and metabolism. Safety monitoring will be performed using scales for side effect, serious adverse events recording, and laboratory tests.

DETAILED DESCRIPTION:
Study design: This study is designed as a randomized, double-blind, placebo-controlled, clinical multi-centre trial. Its main objective is to evaluate the efficacy of SFN vs placebo in decreasing risk and conversion rate of psychosis in CHR population. A total of 300 CHR subjects will be recruited at eight research centres. All participants will be provided withan explanation about the study, and informed consent will be obtained from each participant before participation. The study duration includes an intervention with SFN or placebo for 52 consecutive weeks, and additional 1-year follow-up. The primary outcome is conversion rate of psychosis at the end of follow-up (104 weeks). The secondary outcomes mainly include conversion rate of psychosis at the end of intervention (52 weeks), the severity and the duration of prodromal symptoms, predictive risk of psychosis conversion, neurocognitive functioning and biomarkers of inflammation, oxidative stress and metabolism in peripheral blood. Safety outcomes include side-effects, serious adverse events, laboratory tests, which will be obtained from all participants.

Setting:This study involves eight research centres in China include Shanghai Mental Health Center, Shanghai Xuhui District Mental Health Center, Shanghai Pudong Nanhui Mental Health Center, Suzhou Guangji Hospital, Second Xiangya Hospital of Central South University, Guangzhou Huiai Hospital, Tianjin Anding Hospital, and the First Affiliated Hospital of Zhengzhou University. Shanghai Mental Health Center is the leading centre. Before the trial, standardized training in interview and rating will be provided to all centres equally.

CHR identification: CHR subjects will be identified in the course of face-to-face interviews using the structured interview for prodromal syndromes (SIPS) (Miller et al., 2002; Miller et al., 2003). CHR subjects meet the criteria of prodromal syndromes (COPS) for the attenuated positive symptom syndrome (APSS), brief intermittent psychotic syndrome (BIPS), or genetic risk and deterioration syndrome (GRDS) according to the SIPS. CHR diagnosis will be made by a panel of senior psychiatrists. Severity of CHR subjects' prodromal symptoms will be assessed using the scale of prodromal symptoms (SOPS) (Miller et al., 1999) based on SIPS. In addition, the Positive and Negative Syndrome Scale (PANSS) will be used for rating the severity of psychotic symptoms.

Inclusion criteria:The inclusion criteria of this study are as follows: (a) Subjects meet the criteria of CHR according to SIPS; (b) Subjects will have no history of being medicated with either antipsychotics or mood stabilizers at their first study visit; (c) Age, within the range of 15 to 45 years; (d) Patients and/or their legal guardians for those younger than 18 year old, can understand and sign informed consent, and agree to take the study interventions and complete all visits and examinations.

Exclusion criteria: The exclusion criteria of this study are as follows: (a) A history of schizophrenia or any other psychotic disorders; (b) Severe physical diseases (ie, cardiac and neurologic diseases, brain trauma, liver and kidney diseases, haematopoietic system and immune system dysfunction), or cancer, or other serious complicated diseases; (c) IQ < 70 is assessed by Wechsler Adult Intelligence Scale-Revised in China, or a specific of developmental delay or intellectual disability; (d) Abnormal laboratory test results with clinical significance which will affect the safety of participants as determined by the investigator; (e) A past and/or current abuse of alcohol, amphetamine or any other psychostimulants; (f) Suicidal ideation, plan, or suicidal behaviour in the last 3 months; (g) Clinically significant allergic reaction to broccoli; (h) Pregnancy or preparing for pregnancy, and/or lactation; (i) Participation in another clinical trial within the last 30 days. (j) Other conditions that make the candidate subject unsuitable for this study as determined by the principal investigators (eg, aggressive behaviour, safety concerns, difficulty to complete the follow-up, etc.).

The study will use the following exit/discontinuation criteria: (a) Voluntary discontinuation by the subject who is at any time free to discontinue his or her participation in the study, without prejudice to further assessment and treatment; (b) Severe non-compliance to protocol as judged by the investigator; (c) Subject meets criteria of transition to psychosis; (d) Subject meets exclusion criteria during the intervention (eg, physical diseases, pregnancy, etc.).

Interventions: A total of 300 CHR subjects will be randomly allocated to SFN group (n = 150) or placebo group (n = 150). The intervention duration with SFN or placebo is 52 consecutive weeks. SFN will be delivered as its precursor GR along with a conversion enzyme, myrosinase, which converts GR to SFN in the body. The dosage is six active tablets (411 μmol GR) per day. ZHIYINGUOSU, SFN-producing dietary supplement, is provided at no cost by Shenzhen Fushan Biotech Co., Ltd. (China). The placebo group will be given six placebo tablets per day. Active and placebo tablets are manufactured uniformly with same appearance and similar smell and taste by Shenzhen Fushan Biotech Co., Ltd. (China). Patient compliance will be assessed using Brief Adherence Rating Scale (BARS). The BARS is a brief, pencil-paper, clinician-administered adherence assessment instrument. It consists of four items: three questions and an overall visual analogue rating scale to assess the proportion of doses taken by the patient in the past month (Byerly, Nakonezny, & Rush, 2008). Tablets counting will be conducted monthly for the whole intervention period. After intervention, a 1-year follow-up will be conducted. Temporary use of antipsychotics or anti-depressants is allowed in the whole trial based on the recommendation of the treating clinician, and the information of specific drugs, dosage, treatment period and rationale will be recorded.

Safety: To evaluate the tolerability, we conducted a safety test in over 100 subjects, with the daily dosage is six active tablets. Apart from mild gastrointestinal discomfort, no significant safety or side-effect issues were found in this test.We also found that taking the tablets just after meal reduced the risk of gastrointestinal discomfort. Procedures in the proposed study allow the subject to increase the dosage gradually if the subject experiences significant gastrointestinal discomfort. If the subject experiences a serious adverse event his or her participation can be terminated.

Outcomes: Clinical investigators will collect general information such as gender, age, height, weight, body mass index, demographics and medical history. In addition, vital signs and laboratory tests results will be obtained. These will include body temperature, arterial pulse, blood pressure, heart rate, complete blood cell count, blood electrolytes (K, Na, Cl) and liver and kidney function tests.

The primary outcome is the 2-year conversion rate of psychosis at the end of follow-up (104 weeks). Psychosis conversion is operationally defined according to the criteria of POPS (presence of psychotic symptoms in SIPS/SOPS). Two are required: (a) at least one positive symptom is present at a psychotic level of intensity (rated at level '6' using SOPS); (b) any criterion symptom at sufficient frequency and duration or urgency: the symptom has occurred over a period of 1 month for at least 1 hour per day at a minimum average frequency of 4 days per week, or the symptom is seriously disorganizing or dangerous.

The secondary outcomes include: (a) the 1-year conversion rate of psychosis at the end of intervention period (52 weeks); (b) scores of SOPS; (c) scores of PANSS; (d) the duration of psychotic symptoms; (e) Global Assessment of Functioning; (f) individual predictive risk of psychosis calculated by NAPLS-2 psychosis risk calculator (Carrion et al., 2016) and SHARP psychosis risk calculator (Zhang et al., 2019); (g) scores of MATRICS consensus cognitive battery (MCCB) (Kern et al., 2008; Nuechterlein et al., 2008); (h) the number of participants who receive antipsychotic treatment during the trial; (i) levels of peripheral blood biomarkers of inflammation, oxidative stress and metabolism. Others: (a) Serious adverse events; (b) side-effects of SFN and placebo will be assessed by Systematic Assessment For Treatment Emergent Events (SAFTEE) scale (Levine & Schooler, 1986); (c) Compliance to SFN or placebo assessed using BARS; (d) Usage of antidepressants or other medications; (e) plasma and urinary measures of GR metabolites.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects meet the criteria of CHR according to the Structured Interview for Prodromal Syndromes (SIPS);
2. Subjects will have no history of being medicated with either antipsychotics or mood stabilizers at their first study visit;
3. Age, within the range of 15 to 45 years;
4. Patients and/or their legal guardians for those younger than 18 year old, can understand and sign informed consent, and agree to take the study interventions and complete all visits and examinations.

Exclusion Criteria:

1. A history of schizophrenia or any other psychotic disorders;
2. Severe physical diseases (ie, cardiac and neurologic diseases, brain trauma, liver and kidney diseases, haematopoietic system and immune system dysfunction), or cancer, or other serious complicated diseases;
3. IQ < 70 is assessed by Wechsler Adult Intelligence Scale-Revised in China, or a specific of developmental delay or intellectual disability;
4. Abnormal laboratory test results with clinical significance which will affect the safety of participants as determined by the investigator;
5. A past and/or current abuse of alcohol, amphetamine or any other psychostimulants;
6. Suicidal ideation, plan, or suicidal behaviour in the last 3 months;
7. Clinically significant allergic reaction to broccoli;
8. Pregnancy or preparing for pregnancy, and/or lactation;
9. Participation in another clinical trial within the last 30 days.
10. Other conditions that make the candidate subject unsuitable for this study as determined by the principal investigators (eg, aggressive behaviour, safety concerns, difficulty to complete the follow-up, etc.).

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-07-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year conversion rate of psychosis | 104 weeks
  The proportion of patients are diagnosed with psychosis in each group

SECONDARY OUTCOMES:
1-year conversion rate of psychosis | 52 weeks
  The proportion of patients is diagnosed with psychosis in each group
Severity of prodromal symptoms | 24 weeks, 52 weeks, 104 weeks
  CHR subject's severity of prodromal symptoms is assessed according to the Scale of Prodromal Symptoms (SOPS) based on the SIPS interview
Severity of psychotic symptom | 24 weeks, 52 weeks, 104 weeks
  CHR subject's severity of psychotic symptom is assessed according to the Positive and Negative Syndrome Scale (PANSS)
Function | 24 weeks, 52 weeks, 104 weeks
  CHR subject's overall function is assessed by Global Assessment of Functioning（GAF）
Predictive risk of psychosis | 24 weeks, 52 weeks, 104 weeks
  Predicted risk of psychosis by online psychosis risk calculator.
Neurocognitive functioning | 24 weeks, 52 weeks, 104 weeks
  The MATRICS consensus cognitive battery (MCCB). Original version of the MCCB comprises 10 standardized cognitive measures for seven cognitive domains: speed of processing, attention/vigilance, working memory (verbal and nonverbal), verbal learning, visual learning, reasoning and problem solving, and social cognition. The 7 domain scores and a composite score were used as variables of neurocognition.Our group has previously contributed to the Chinese norms for the MCCB scores of tests. The kappa values for test-retest reliability of the subtests of the Chinese version ranges from 0.73 to 0.94.
Level of inflammation in subjects' peripheral blood | 24 weeks, 52 weeks, 104 weeks
  Detecting expression levels of inflammation-related biomarkers in peripheral blood.
Level of oxidative stress in subjects' peripheral blood | 24 weeks, 52 weeks, 104 weeks
  Detecting expression levels of oxidative stress-related biomarkers in peripheral blood.
Level of metabolism in subjects' peripheral blood | 24 weeks, 52 weeks, 104 weeks
  Detecting expression levels of metabolism-related biomarkers in peripheral blood.

OTHER OUTCOMES:
Serious adverse events | the whole process
  Serious adverse events
Side-effects of SFN and placebo | 52 weeks
  side-effects of SFN and placebo will be assessed by Systematic Assessment For Treatment Emergent Events (SAFTEE) scale
Compliance | 24 weeks
  Compliance to SFN or placebo assessed using Brief Adherence Rating Scale
Number of CHR subjects who use antidepressants or other medications | 52 weeks
  Usage of antidepressants or other medications
Plasma and urinary measures of GR metabolites | 24 weeks, 52 weeks, 104 weeks
  Plasma and urinary measures of GR metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Jijun Wang, PhD, Study Director — Shanghai Mental Health Center; Tianhong Zhang, PhD, Principal Investigator — Shanghai Mental Health Center; Hua Jin, PhD, Principal Investigator — University of California, San Diego; Xiaolong Li, PhD, Principal Investigator — Shenzhen Fushan Biotech Co., Ltd.
Locations (9):
- China (9):
  - Guangzhou Psychiatric Hospital, Guangzhou, Guangdong
  - the First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Suzhou Psychiatric Hospital, Suzhou, Jiangsu
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - Shanghai Xuhui District Mental Health Center, Shanghai, Shanghai Municipality
  - Shanghai Pudong Nanhui Mental Health Center, Shanghai, Shanghai Municipality
  - Shenzhen Kangning Hospital, Shenzhen, Shenzhen
  - Tianjin Anding Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Miller TJ, McGlashan TH, Rosen JL, Cadenhead K, Cannon T, Ventura J, McFarlane W, Perkins DO, Pearlson GD, Woods SW. Prodromal assessment with the structured interview for prodromal syndromes and the scale of prodromal symptoms: predictive validity, interrater reliability, and training to reliability. Schizophr Bull. 2003;29(4):703-15. doi: 10.1093/oxfordjournals.schbul.a007040. PMID 14989408
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] Carrion RE, Cornblatt BA, Burton CZ, Tso IF, Auther AM, Adelsheim S, Calkins R, Carter CS, Niendam T, Sale TG, Taylor SF, McFarlane WR. Personalized Prediction of Psychosis: External Validation of the NAPLS-2 Psychosis Risk Calculator With the EDIPPP Project. Am J Psychiatry. 2016 Oct 1;173(10):989-996. doi: 10.1176/appi.ajp.2016.15121565. Epub 2016 Jul 1. PMID 27363511
- [Background] Zhang T, Xu L, Tang Y, Li H, Tang X, Cui H, Wei Y, Wang Y, Hu Q, Liu X, Li C, Lu Z, McCarley RW, Seidman LJ, Wang J; SHARP (ShangHai At Risk for Psychosis) Study Group. Prediction of psychosis in prodrome: development and validation of a simple, personalized risk calculator. Psychol Med. 2019 Sep;49(12):1990-1998. doi: 10.1017/S0033291718002738. Epub 2018 Sep 14. PMID 30213278
- [Background] Nuechterlein KH, Green MF, Kern RS, Baade LE, Barch DM, Cohen JD, Essock S, Fenton WS, Frese FJ 3rd, Gold JM, Goldberg T, Heaton RK, Keefe RS, Kraemer H, Mesholam-Gately R, Seidman LJ, Stover E, Weinberger DR, Young AS, Zalcman S, Marder SR. The MATRICS Consensus Cognitive Battery, part 1: test selection, reliability, and validity. Am J Psychiatry. 2008 Feb;165(2):203-13. doi: 10.1176/appi.ajp.2007.07010042. Epub 2008 Jan 2. PMID 18172019
- [Background] Kern RS, Nuechterlein KH, Green MF, Baade LE, Fenton WS, Gold JM, Keefe RS, Mesholam-Gately R, Mintz J, Seidman LJ, Stover E, Marder SR. The MATRICS Consensus Cognitive Battery, part 2: co-norming and standardization. Am J Psychiatry. 2008 Feb;165(2):214-20. doi: 10.1176/appi.ajp.2007.07010043. Epub 2008 Jan 2. PMID 18172018
- [Background] Addington J, Liu L, Buchy L, Cadenhead KS, Cannon TD, Cornblatt BA, Perkins DO, Seidman LJ, Tsuang MT, Walker EF, Woods SW, Bearden CE, Mathalon DH, McGlashan TH. North American Prodrome Longitudinal Study (NAPLS 2): The Prodromal Symptoms. J Nerv Ment Dis. 2015 May;203(5):328-35. doi: 10.1097/NMD.0000000000000290. PMID 25919383
- [Background] Li H, Zhang T, Xu L, Tang Y, Cui H, Wei Y, Tang X, Woodberry KA, Shapiro DI, Li C, Seidman LJ, Wang J. A comparison of conversion rates, clinical profiles and predictors of outcomes in two independent samples of individuals at clinical high risk for psychosis in China. Schizophr Res. 2018 Jul;197:509-515. doi: 10.1016/j.schres.2017.11.029. Epub 2017 Dec 26. PMID 29287626
- [Background] Singh K, Connors SL, Macklin EA, Smith KD, Fahey JW, Talalay P, Zimmerman AW. Sulforaphane treatment of autism spectrum disorder (ASD). Proc Natl Acad Sci U S A. 2014 Oct 28;111(43):15550-5. doi: 10.1073/pnas.1416940111. Epub 2014 Oct 13. PMID 25313065
- [Background] Bent S, Lawton B, Warren T, Widjaja F, Dang K, Fahey JW, Cornblatt B, Kinchen JM, Delucchi K, Hendren RL. Identification of urinary metabolites that correlate with clinical improvements in children with autism treated with sulforaphane from broccoli. Mol Autism. 2018 May 30;9:35. doi: 10.1186/s13229-018-0218-4. eCollection 2018. PMID 29854372
- [Background] Li Z, Zhang T, Xu L, Wei Y, Tang Y, Hu Q, Liu X, Li X, Davis J, Smith R, Jin H, Wang J. Decreasing risk of psychosis by sulforaphane study protocol for a randomized, double-blind, placebo-controlled, clinical multi-centre trial. Early Interv Psychiatry. 2021 Jun;15(3):585-594. doi: 10.1111/eip.12988. Epub 2020 May 21. PMID 32436318